CLINICAL TRIAL: NCT01444027
Title: A Problem Solving Intervention for Hospice Caregivers
Brief Title: Hospice Problem Solving Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, George Demiris, Professor, Biobehavioral Nursing and Health Systems, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 36909; 1R01NR012213-01A1 (NIH)
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Hospice Informal Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Attention Control (No Intervention): This group receives standard care with the attention of social support/ "friendly interactions" and serves as an attention control group.
- Intervention Group 1 (Face to Face) (Experimental): This group receives Problem Solving Therapy in face to face visits.
  Interventions: Behavioral: Problem Solving Therapy
- Intervention Group 2 (Video) (Experimental): This group receives Problem Solving Therapy via video.
  Interventions: Behavioral: Problem Solving Therapy

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem-solving therapy (PST) focuses on behavioral change principles derived from this theoretical framework. PST addresses four skills: 1) problem definition and formulation, which involves gathering data and information, articulating the issue in clear terms, identifying the challenge, and setting realistic goals; 2) generation of alternative strategies; 3) decision making; and 4) solution implementation. The intervention is delivered in a series of interactions with the interventionist.
  Arms: Intervention Group 1 (Face to Face); Intervention Group 2 (Video)

SUMMARY:
In recent years, the demand for home hospice care has grown rapidly. Family members and friends who act as informal caregivers are essential to the provision of palliative care services; however, this role is not without adverse effects on the caregivers themselves. It is well documented that emotional needs of individuals caring for dying persons in their home are not well attended, and interventions aiming to provide support to informal hospice caregivers are notably lacking. In this context, problem solving therapy (PST) provides an overall coping process that fosters adaptive situational coping and behavioral competence. The investigators are conducting a randomized controlled trial to fully evaluate the PST intervention for informal hospice caregivers. Additionally, the investigators aim to evaluate how the modality of the intervention (face to face vs video) impacts its effectiveness. This investigator team is conducting a 4-year randomized trial study in which hospice caregivers will be randomly assigned to a group receiving standard hospice care with the addition of social support interactions (attention control group) or a group receiving standard hospice care with the addition of the problem solving intervention delivered face to face (intervention group 1) or a group receiving standard hospice care with the addition of the problem solving intervention delivered via video (intervention group 2). The specific aims include an assessment of the impact of PST on caregiver quality of life, problem solving ability, and caregiver anxiety.

ELIGIBILITY:
Inclusion Criteria:

* enrolled as a family/informal caregiver of a hospice patient
* 18 years or older
* with access to a standard phone line or Internet and computer access at home
* without functional hearing loss or with a hearing aid that allows the participant to conduct telephone conversations as assessed by the research staff (by questioning and observing the caregiver)
* no or only mild cognitive impairment
* speak and read English, with at least a 6th-grade education

Exclusion Criteria:

* lack of phone or Internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2011-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Demiris, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Starr LT, Bullock K, Washington K, Aryal S, Parker Oliver D, Demiris G. Anxiety, Depression, Quality of Life, Caregiver Burden, and Perceptions of Caregiver-Centered Communication among Black and White Hospice Family Caregivers. J Palliat Med. 2022 Apr;25(4):596-605. doi: 10.1089/jpm.2021.0302. Epub 2021 Nov 18. PMID 34793244
- [Derived] Demiris G, Oliver DP, Washington K, Pike K. A Problem-Solving Intervention for Hospice Family Caregivers: A Randomized Clinical Trial. J Am Geriatr Soc. 2019 Jul;67(7):1345-1352. doi: 10.1111/jgs.15894. Epub 2019 Apr 4. PMID 30946495
- [Derived] Benson JJ, Parker Oliver D, Demiris G, Washington K. Accounts of Family Conflict in Home Hospice Care: The Central Role of Autonomy for Informal Caregiver Resilience. J Fam Nurs. 2019 May;25(2):190-218. doi: 10.1177/1074840719828091. Epub 2019 Feb 17. PMID 30773970
- [Derived] Tarter R, Demiris G, Pike K, Washington K, Parker Oliver D. Pain in Hospice Patients With Dementia: The Informal Caregiver Experience. Am J Alzheimers Dis Other Demen. 2016 Sep;31(6):524-9. doi: 10.1177/1533317516653825. Epub 2016 Jun 14. PMID 27303062
- [Derived] Oliver DP, Demiris G, Washington KT, Clark C, Thomas-Jones D. Challenges and Strategies for Hospice Caregivers: A Qualitative Analysis. Gerontologist. 2017 Aug 1;57(4):648-656. doi: 10.1093/geront/gnw054. PMID 27048707
- [Derived] Washington KT, Pike KC, Demiris G, Parker Oliver D, Albright DL, Lewis AM. Gender Differences in Caregiving at End of Life: Implications for Hospice Teams. J Palliat Med. 2015 Dec;18(12):1048-53. doi: 10.1089/jpm.2015.0214. Epub 2015 Oct 20. PMID 26484426
- [Derived] Washington KT, Pike KC, Demiris G, Oliver DP. Unique characteristics of informal hospice cancer caregiving. Support Care Cancer. 2015 Jul;23(7):2121-8. doi: 10.1007/s00520-014-2570-z. Epub 2014 Dec 30. PMID 25547480
- [Derived] Washington KT, Wittenberg-Lyles E, Oliver DP, Baldwin PK, Tappana J, Wright JH, Demiris G. Rethinking family caregiving: tailoring cognitive-behavioral therapies to the hospice experience. Health Soc Work. 2014 Nov;39(4):244-50. doi: 10.1093/hsw/hlu031. PMID 25369725
- [Derived] Washington KT, Demiris G, Pike KC, Kruse RL, Oliver DP. Anxiety among informal hospice caregivers: an exploratory study. Palliat Support Care. 2015 Jun;13(3):567-73. doi: 10.1017/S1478951513001193. Epub 2014 Feb 13. PMID 24524662
- [Derived] Demiris G, Parker Oliver D, Capurro D, Wittenberg-Lyles E. Implementation science: implications for intervention research in hospice and palliative care. Gerontologist. 2014 Apr;54(2):163-71. doi: 10.1093/geront/gnt022. Epub 2013 Apr 4. PMID 23558847

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
Started | 172 | 171 | 171
Received Intervention as Assigned | 168 | 161 | 147
1 Month Follow-up | 160 | 159 | 141
3 Month Follow-up | 142 | 141 | 133
Completed | 142 | 141 | 133
Not Completed | 30 | 30 | 38
Not completed — Withdrawal by Subject | 4 | 10 | 24
Not completed — Lost to Follow-up | 26 | 20 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video) | Total
Number analyzed (Participants) | 172 | 171 | 171 | 514
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (13.6) | 59.9 (11.6) | 61.3 (12.0) | 60.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 125 | 129 | 386
  Male | 40 | 46 | 42 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 4
  Asian | 9 | 8 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 8 | 5 | 16
  White | 155 | 153 | 152 | 460
  More than one race | 4 | 1 | 5 | 10
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 172 | 171 | 171 | 514

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Anxiety: Change From Baseline to Post-Intervention Exit
Description: Caregiver anxiety was measured with the 7-item Generalized Anxiety Disorder (GAD-7) Scale (Spitzer et al., 2006), which measures the frequency with which respondents experience symptoms of anxiety such as restlessness, difficulty relaxing, and uncontrollable worrying. The GAD-7 total scores range from 0 to 21, with higher scores indicating more anxiety.
Time Frame: At Baseline and Exit (approximately 4 weeks after recruitment)
Population: Intent to treat population (all participants who received at least one intervention session). Multiple imputation was used to replace missing data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
Number analyzed (Participants) | 172 | 171 | 171
units on a scale | -0.9 (0.3) | -2.0 (0.4) | -0.7 (0.4)
Statistical Analysis 1: Comparison: Attention Control vs Intervention Group 1 (Face to Face); Test type: Superiority; p = 0.002, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 2: Comparison: Attention Control vs Intervention Group 2 (Video); Test type: Superiority; p = 0.90, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons
Statistical Analysis 3: Comparison: Intervention Group 1 (Face to Face) vs Intervention Group 2 (Video); Test type: Superiority; p = 0.002, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status

2. Primary Outcome: Caregiver Quality of Life - Physical: Change From Baseline to Post-Intervention Exit
Description: An interview CQLI version was developed by using identical items from the paper-based CQLI and replacing the visual analogue response format with a 0-10 response scale. Higher scores indicate better physical quality of life.
Time Frame: At Baseline and Exit (approximately 4 weeks after recruitment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
Number analyzed (Participants) | 172 | 171 | 171
units on a scale | -0.4 (0.1) | 0.2 (0.1) | -0.2 (0.1)
Statistical Analysis 1: Comparison: Attention Control vs Intervention Group 1 (Face to Face); Test type: Superiority; p = 0.001, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for the baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 2: Comparison: Attention Control vs Intervention Group 2 (Video); Test type: Superiority; p = 0.48, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 3: Comparison: Intervention Group 1 (Face to Face) vs Intervention Group 2 (Video); Test type: Superiority; p = .01, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status

3. Primary Outcome: Caregiver Quality of Life - Social: Change From Baseline to Post-Intervention Exit
Description: An interview CQLI version was developed by using identical items from the paper-based CQLI and replacing the visual analogue response format with a 0-10 response scale. Higher scores indicate better social quality of life.
Time Frame: At Baseline and Exit (approximately 4 weeks after recruitment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
Number analyzed (Participants) | 172 | 171 | 171
units on a scale | -0.2 (0.2) | 0.2 (0.1) | -0.4 (0.2)
Statistical Analysis 1: Comparison: Attention Control vs Intervention Group 1 (Face to Face); Test type: Superiority; p = 0.001, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 2: Comparison: Attention Control vs Intervention Group 2 (Video); Test type: Superiority; p = 0.83, Regression, Linear; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 3: Comparison: Intervention Group 1 (Face to Face) vs Intervention Group 2 (Video); Test type: Superiority; p = 0.001, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status

4. Primary Outcome: Caregiver Quality of Life - Emotional: Change From Baseline to Post-Intervention Exit
Description: An interview CQLI version was developed by using identical items from the paper-based CQLI and replacing the visual analogue response format with a 0-10 response scale. Higher scores indicate better emotional quality of life.
Time Frame: At Baseline and Exit (approximately 4 weeks after recruitment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
Number analyzed (Participants) | 172 | 171 | 171
units on a scale | -0.1 (0.2) | 0.4 (0.1) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Attention Control vs Intervention Group 1 (Face to Face); Test type: Superiority; p = 0.003, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 2: Comparison: Attention Control vs Intervention Group 2 (Video); Test type: Superiority; p = 0.16, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 3: Comparison: Intervention Group 1 (Face to Face) vs Intervention Group 2 (Video); Test type: Superiority; p = 0.17, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status

5. Primary Outcome: Caregiver Quality of Life - Financial: Change From Baseline to Post-Intervention Exit
Description: An interview CQLI version was developed by using identical items from the paper-based CQLI and replacing the visual analogue response format with a 0-10 response scale. Higher scores indicate better financial quality of life.
Time Frame: At Baseline and Exit (approximately 4 weeks after recruitment)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
Number analyzed (Participants) | 172 | 171 | 171
units on a scale | 0.0 (0.1) | 0.5 (0.1) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Attention Control vs Intervention Group 1 (Face to Face); Test type: Superiority; p = 0.001, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 2: Comparison: Attention Control vs Intervention Group 2 (Video); Test type: Superiority; p = 0.78, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status
Statistical Analysis 3: Comparison: Intervention Group 1 (Face to Face) vs Intervention Group 2 (Video); Test type: Superiority; p = 0.004, Regression, Linear — Bonferroni adjusted p-value for 3 pairwise comparisons; Adjusted for baseline value of the measure, hospice agency, and bereaved status

ADVERSE EVENTS:
Time Frame: 3 months
Description: Caregivers are participants in this study and all cause mortality is reported for them, not their loved one receiving hospice care
Arm/Group | Attention Control | Intervention Group 1 (Face to Face) | Intervention Group 2 (Video)
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/171 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/172 | 0/171 | 0/272
Other Adverse Events (participants affected / at risk) | 0/172 | 0/171 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No